CLINICAL TRIAL: NCT00581451
Title: A 3-Part, Randomized, Multiple-Dose, Sequential Design Study of Bifeprunox in Healthy Subjects in Order to Establish a Titration Regimen With an Improved Tolerability Profile
Brief Title: Study Evaluating the Tolerability of Bifeprunox in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: 3168A2-1005
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
MeSH Terms: interventions — bifeprunox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): bifeprunox 25 day
  Interventions: Drug: bifeprunox
- B (Experimental): bifeprunox 14 day
  Interventions: Drug: bifeprunox
- C (Experimental): bifeprunox 14 day
  Interventions: Drug: bifeprunox
- D (Experimental): bifeprunox 9 day
  Interventions: Drug: bifeprunox

INTERVENTIONS:
Drug: bifeprunox — oral tablet once daily

SUMMARY:
Safety and tolerability study in healthy volunteers

ELIGIBILITY:
Inclusion criteria:

* Healthy male 18-50 years
* Nonlactating female 18-50 years

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Tolerability | 28 days

SECONDARY OUTCOMES:
Safety | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer